CLINICAL TRIAL: NCT00157040
Title: Recombinant Antihemophilic Factor (rAHF-PFM) Manufactured and Formulated Without Added Human or Animal Proteins: Evaluation of Pharmacokinetics, Immunogenicity, Efficacy and Safety in Previously Treated Pediatric Patients With Hemophilia A
Brief Title: Study of Pharmacokinetics, Efficacy, and Safety of a Recombinant and Protein-Free Factor VIII (rAHF-PFM) in Pediatric Patients With Hemophilia A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060101
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
Keywords: Factor VIII Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

INTERVENTIONS:
Drug: Antihemophilic factor, recombinant, manufactured protein-free

SUMMARY:
The purpose of this study is to evaluate whether rAHF-PFM is effective and safe in the treatment of children with hemophilia A. The study consists of 2 parts. Part 1 of the study is a pharmacokinetic evaluation, and Part 2 is an evaluation of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject is less than 6 years of age
* Severe or moderately-severe hemophilia A as defined by a baseline factor VIII level <= 2%, documented at screening or on the basis of historical data (e.g., at hemophilia diagnosis)
* Documented medical history of at least 50 exposure days for treatment with all other factor VIII products
* Subject's parent or legally authorized representative has provided informed consent

Exclusion Criteria:

* Detectable inhibitor to factor VIII measured in the screening sample by the local or central hemostasis laboratory
* History of inhibitor to factor VIII at any time prior to screening
* Subject has any one of the following laboratory abnormalities at the time of screening:

  1. platelet count < 100,000/mm3
  2. hemoglobin concentration < 10 g/dL (100 g/L)
  3. serum creatinine > 1.5 times the ULN for age
  4. total bilirubin > 2 times the ULN for age
* Subject has an inherited or acquired hemostatic defect other than hemophilia A (e.g., platelet dysfunction secondary to uremia, liver failure, von Willebrand's Disease)
* Subject has known hypersensitivity to RECOMBINATE rAHF
* Subject is currently participating in another investigational drug study or has participated in any clinical study involving an investigational drug within 30 days of study entry
* Subject is identified by the investigator as being unable or unwilling to cooperate with study procedures

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2002-06-07 (Actual); Primary Completion 2005-01-04 (Actual); Study Completion 2005-01-04 (Actual)

PRIMARY OUTCOMES:
The terminal phase half-life of Recombinant Antihemophilic Factor (rAHF-PFM) | Within 30 minutes prior to the pharmacokinetic infusion and at 1 hour ± 5 minutes, 9 ± 1 hour, 24 ± 2 hours, and 48 ± 2 hours after the infusion
  Terminal phase half-life of rAHF-PFM was to be determined using the biphasic linear regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (10):
  - Children´s Hospital Los Angeles, Los Angeles, California
  - Emory University, Department of Pediatrics, Atlanta, Georgia
  - Children´s Memorial Hospital, Chicago, Illinois
  - Comprehensive Bleeding Disorders Center, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa Regional Hemophilia Center, Department of Pediatrics, Iowa City, Iowa
  - University of Michigan Hemophilia Treatment Center, Ann Arbor, Michigan
  - Children´s Hospital of Michigan, Detroit, Michigan
  - Children´s Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Health Science Center, Houston, Texas
- Hospital for Sick Children, Division of Hematology/Oncology, Toronto, Ontario, Canada
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Shapiro A, Gruppo R, Pabinger I, Collins PW, Hay CR, Schroth P, Casey K, Patrone L, Ehrlich H, Ewenstein BM. Integrated analysis of safety and efficacy of a plasma- and albumin-free recombinant factor VIII (rAHF-PFM) from six clinical studies in patients with hemophilia A. Expert Opin Biol Ther. 2009 Mar;9(3):273-83. doi: 10.1517/14712590902729392. PMID 19216617